CLINICAL TRIAL: NCT03130959
Title: Phase Ib /II Clinical Trial of Nivolumab Monotherapy and Nivolumab in Combination With Ipilimumab in Pediatric Subjects With High Grade Primary CNS Malignancies
Brief Title: A Study to Evaluate the Safety and Efficacy of Nivolumab Monotherapy and Nivolumab in Combination With Ipilimumab in Pediatric Participants With High Grade Primary Central Nervous System (CNS) Malignancies
Acronym: CheckMate 908
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-908; 2016-004441-82 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2017-04-05; First posted 2017-04-27 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module A (Experimental)
  Interventions: Biological: Nivolumab
- Module B (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo, BMS-936558
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy, BMS-734016
  Arms: Module B

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of nivolumab alone and in combination with ipilimumab in pediatric patients with high grade primary central nervous system (CNS) malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Must have received standard of care therapy, and there must be no potentially-curative treatment available, in one of the following cohorts:
* A newly diagnosed Diffuse Intrinsic Pontine Glioma (DIPG) that has been treated with radiation therapy (RT) but no chemotherapy
* A histologically confirmed recurrent or progressive non-brainstem High Grade Glioma (HGG) previously treated with surgical resection and RT
* A histologically confirmed medulloblastoma that has relapsed or is resistant to at least one line of prior therapy including surgery, RT, and chemotherapy
* A histologically confirmed ependymoma that has relapsed or is resistant to at least one line of prior therapy including surgical resection and RT
* A histologically-confirmed high grade CNS malignancy "other than above" which is recurrent or progressive after at least one line of prior therapy
* Lansky play score (LPS) for ≤ 16 years of age or Karnofsky performance scale (KPS) for > 16 years of age assessed within two weeks of enrollment must be >= 60
* A tumor sample must be available for submission to central laboratory (not required for DIPG)

Exclusion Criteria:

* An active, known, or suspected autoimmune disease
* A concurrent condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of start of study treatment
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Other protocol defined inclusion/exclusion criteria apply

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (54):
- United States (14):
  - Local Institution - 0057, Los Angeles, California
  - Local Institution - 0016, Aurora, Colorado
  - Local Institution - 0046, Gainesville, Florida
  - Local Institution - 0011, Chicago, Illinois
  - Local Institution - 0005, Baltimore, Maryland
  - Local Institution - 0043, Boston, Massachusetts
  - Local Institution - 0044, St Louis, Missouri
  - Local Institution - 0004, New York, New York
  - Local Institution - 0017, New York, New York
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - Local Institution - 0066, Philadelphia, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution - 0012, Memphis, Tennessee
  - Local Institution - 0042, Houston, Texas
- Australia (5):
  - Local Institution - 0022, Randwick, New South Wales
  - Local Institution - 0035, Sth Brisbane, Queensland
  - Local Institution, Clayton, Victoria
  - Local Institution - 0034, Parkville, Victoria
  - Local Institution - 0033, Nedlands, Western Australia
- Brazil (5):
  - Local Institution - 0052, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0051, Barretos, São Paulo
  - Local Institution - 0053, Ribeirão Preto, São Paulo
  - Local Institution - 0049, São Paulo
  - Local Institution - 0050, São Paulo
- Canada (3):
  - Local Institution - 0021, Toronto, Ontario
  - Local Institution - 0001, Montreal, Quebec
  - Local Institution - 0002, Québec, Quebec
- France (8):
  - Local Institution - 0028, Angers
  - Local Institution - 0029, Bordeaux
  - Local Institution - 0027, Lille
  - Local Institution - 0025, Lyon
  - Local Institution - 0024, Marseille
  - Local Institution - 0023, Paris
  - Local Institution - 0064, Vandœuvre-lès-Nancy
  - Local Institution - 0026, VIillejuif
- Germany (4):
  - Local Institution - 0060, Essen
  - Local Institution - 0061, Hamburg
  - Local Institution - 0063, Heidelberg
  - Local Institution - 0062, Würzburg
- Local Institution - 0018, Hong Kong, Hong Kong
- Israel (2):
  - Local Institution - 0059, Haifa
  - Local Institution - 0058, Ramat Gan
- Netherlands (2):
  - Local Institution - 0007, Rotterdam
  - Local Institution - 0008, Utrecht
- Local Institution - 0067, Oslo, Norway
- Local Institution - 0047, Warsaw, Poland
- Local Institution - 0048, Moscow, Russia
- Spain (3):
  - Local Institution - 0037, Esplugues de Llobregat
  - Local Institution - 0038, Madrid
  - Local Institution - 0036, Valencia
- Local Institution - 0065, Solna, Sweden
- United Kingdom (3):
  - Local Institution - 0010, London, Greater London
  - Local Institution - 0013, Liverpool, Merseyside
  - Local Institution - 0015, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunkel IJ, Doz F, Foreman NK, Hargrave D, Lassaletta A, Andre N, Hansford JR, Hassall T, Eyrich M, Gururangan S, Bartels U, Gajjar A, Howell L, Warad D, Pacius M, Tam R, Wang Y, Zhu L, Cohen K. Nivolumab with or without ipilimumab in pediatric patients with high-grade CNS malignancies: Safety, efficacy, biomarker, and pharmacokinetics-CheckMate 908. Neuro Oncol. 2023 Aug 3;25(8):1530-1545. doi: 10.1093/neuonc/noad031. PMID 36808285
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 participants were treated
Groups:
- Arm A1: Module A: nivolumab 3 mg/kg every 2 weeks.
  Cohort 1: participants with newly-diagnosed DIPG, including midline glioma with H3K27M mutation.
- Arm B1: Module B: nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks, for 4 doses, then nivolumab 3 mg/kg every 2 weeks thereafter.
  Cohort 1: participants with newly-diagnosed DIPG, including midline glioma with H3K27M mutation.
- Arm A2: Module A: nivolumab 3 mg/kg every 2 weeks.
  Cohort 2: participants with recurrent or progressive non-brainstem HGG, regardless of mutation status, including glioblastoma.
- Arm B2: Module B: nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks, for 4 doses, then nivolumab 3 mg/kg every 2 weeks thereafter.
  Cohort 2: participants with recurrent or progressive non-brainstem HGG, regardless of mutation status, including glioblastoma.
- Arm A3: Module A: nivolumab 3 mg/kg every 2 weeks.
  Cohort 3: participants with relapsed or resistant medulloblastoma.
- Arm B3: Module B: nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks, for 4 doses, then nivolumab 3 mg/kg every 2 weeks thereafter.
  Cohort 3: participants with relapsed or resistant medulloblastoma.
- Arm A4: Module A: nivolumab 3 mg/kg every 2 weeks.
  Cohort 4: participants with relapsed or resistant ependymoma.
- Arm B4: Module B: nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks, for 4 doses, then nivolumab 3 mg/kg every 2 weeks thereafter.
  Cohort 4: participants with relapsed or resistant ependymoma.
- Arm A5: Module A: nivolumab 3 mg/kg every 2 weeks.
  Cohort 5: participants with other recurrent subtypes of high-grade CNS malignancy (eg, pineoblastoma, AT/RT, germ cell tumor, and others).
- Arm B5: Module B: nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks, for 4 doses, then nivolumab 3 mg/kg every 2 weeks thereafter.
  Cohort 5: participants with other recurrent subtypes of high-grade CNS malignancy (eg, pineoblastoma, AT/RT, germ cell tumor, and others).
Period: Overall Study
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Started (Started = initiated treatment) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Completed (Completed = completed treatment) | 0 | 12 | 0 | 1 | 0 | 9 | 0 | 6 | 0 | 4
Not Completed | 23 | 10 | 16 | 14 | 15 | 6 | 12 | 4 | 19 | 15
Not completed — Disease progression | 19 | 7 | 12 | 7 | 12 | 3 | 6 | 3 | 15 | 8
Not completed — Study drug toxicity | 2 | 2 | 1 | 2 | 1 | 1 | 3 | 0 | 3 | 3
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Subject request to discontinue therapy | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Not reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event unrelated to drug | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Participant withdrew consent | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Administrative reason by sponsor | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5 | Total
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19 | 166
Age, Customized [Count of Participants; unit: Participants]
  < 2 years old | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  >= 2 and < 12 years old | 15 | 16 | 6 | 5 | 4 | 4 | 8 | 4 | 13 | 12 | 87
  >= 12 and < 18 years old | 6 | 5 | 6 | 8 | 11 | 9 | 3 | 3 | 4 | 6 | 61
  >= 18 years old | 2 | 1 | 4 | 2 | 0 | 2 | 1 | 2 | 1 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 6 | 3 | 5 | 5 | 6 | 3 | 4 | 10 | 70
  Male | 11 | 6 | 10 | 12 | 10 | 10 | 6 | 7 | 15 | 9 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 14
  Not Hispanic or Latino | 7 | 10 | 4 | 5 | 6 | 4 | 5 | 5 | 8 | 6 | 60
  Unknown or Not Reported | 14 | 9 | 10 | 8 | 9 | 10 | 6 | 4 | 9 | 13 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 11 | 13 | 14 | 14 | 14 | 7 | 9 | 18 | 13 | 132
  Black or African American | 2 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 9
  Asian | 0 | 2 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 10
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 2 | 4 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Safety Lead-In Participants With Dose Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) is defined as a drug-related AE occurring in the first 6 weeks of study treatment. A participant was considered evaluable for a DLT if study treatment was delayed > 2 weeks or was discontinued due to a related Adverse Event (AE), or if planned study treatment (3 doses of nivolumab in Module A, 2 doses of nivolumab plus ipilimumab in Module B) was administered and safety evaluation after 6 weeks on study is available to the study steering committee (SSC).
Time Frame: up to 6 weeks post-dosing
Population: Safety Lead-in participants: In Module A, the first 6 DLT-evaluable participants in Cohort 1 and the first 10 DLT-evaluable participants in Cohorts 2-5; in Module B, the first 10 DLT-evaluable participants.
Measure: Number; unit: Number of participants
Groups:
- Arm A1, Safety Lead-in: Module A, Cohort 1
- Arms A2-A5, Safety Lead-in: Module A, Cohorts 2 through 5
- Arms B2-B5, Safety Lead-in: Module B, Cohorts 2 through 5
Arm/Group | Arm A1, Safety Lead-in | Arms A2-A5, Safety Lead-in | Arms B2-B5, Safety Lead-in
Number analyzed (Participants) | 15 | 10 | 16
Number of participants | 0 | 0 | 0

2. Primary Outcome: Number of Safety Lead-In Participants With Serious Adverse Events (SAEs)
Description: The number of Safety Lead-In Participants who experienced a Serious Adverse Event (SAE) during the course of the study.
Time Frame: up to 6 weeks post-dosing
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Arm A1, Safety Lead-in | Arms A2-A5, Safety Lead-in | Arms B2-B5, Safety Lead-in
Number analyzed (Participants) | 15 | 10 | 16
Number of participants | 7 | 6 | 8

3. Primary Outcome: Number of Safety Lead-In Participants With Adverse Events (AEs) Leading to Discontinuation
Description: The number of Safety Lead-In Participants who experienced an Adverse Event (AE) during the course of the study that lead to discontinuation of study therapy.
Time Frame: From first dose to 30 days post-last dose (up to approximately 6 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1, Safety Lead-in | Arms A2-A5, Safety Lead-in | Arms B2-B5, Safety Lead-in
Number analyzed (Participants) | 15 | 10 | 16
Participants | 3 | 4 | 2

4. Primary Outcome: Overall Survival (OS), Cohort 1 Only
Description: Overall survival (OS) is defined as the time between the date of diagnosis and the date of death in Cohort 1.
Time Frame: up to approximately 42 months
Population: All treated participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Arm A1 | Arm B1
Number analyzed (Participants) | 23 | 22
months | 11.66 [10.32 to 16.46] | 10.78 [9.13 to 15.77]

5. Primary Outcome: Progression-Free Survival (PFS), Cohorts 2-4
Description: Progression-free survival (PFS) is defined as the time from first dose to the date of the first documented tumor progression or death due to any cause.
Time Frame: up to approximately 42 months
Population: All treated participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 12 | 10
months | 1.74 [1.35 to 2.73] | 1.31 [1.18 to 1.45] | 1.38 [1.22 to 1.38] | 2.76 [1.48 to 4.53] | 1.41 [1.41 to 2.60] | 4.60 [1.41 to 5.39]

6. Primary Outcome: Progression-Free Survival (PFS), Cohort 5 Only
Description: as for outcome 5
Time Frame: up to approximately 42 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A5 | Arm B5
Number analyzed (Participants) | 19 | 19
months | 1.22 [1.08 to 1.31] | 1.61 [1.31 to 3.45]

7. Secondary Outcome: Progression-Free Survival (PFS), Cohort 1 Only
Description: Progression-free survival (PFS) is defined as the time from first dose to the date of the first documented tumor progression or death due to any cause.
  Progression is defined as:
  * ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement
  * Significant increase in T2 or fast fluid-attenuated inversion recovery (FLAIR) non-enhancing lesions on stable or increasing doses of corticosteroids
  * Any new lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor
  * Failure to return for evaluation as a result of death or deteriorating condition
  * Clear progression of non-measurable disease
Time Frame: From first dose to the date of the first documented tumor progression or death due to any cause (up to approximately 55 months)
Population: All treated participants in Cohort 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm B1
Number analyzed (Participants) | 23 | 22
Months | 6.21 [3.75 to 6.54] | 4.53 [2.99 to 6.44]

8. Secondary Outcome: Overall Survival at 12 Months (OS12), Cohorts 1-4
Description: Overall survival at 12 months (OS12) is defined as the percentage of participants who are alive at 12 months, measured as the survival rate at 12 months from Kaplan-Meier product limit cumulative probability.
Time Frame: From first dose to up to 12 months after first dose
Population: All treated participants in Cohorts 1-4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10
Percentage of participants | 47.3 [25.2 to 66.5] | 42.9 [21.9 to 62.3] | 37.5 [15.4 to 59.8] | 32.8 [10.5 to 57.6] | 38.9 [14.3 to 63.2] | 86.7 [56.4 to 96.5] | 41.7 [15.2 to 66.5] | 44.4 [13.6 to 71.9]

9. Secondary Outcome: Progression-Free Survival at 6 Months (PFS6), Cohorts 2-5
Description: Progression-free survival at 6 months (PFS6) is defined as the percentage of participants who are progression free and alive at 6 months following first dose date, measured as the survival rate at 6 months from Kaplan-Meier product limit cumulative probability of progression free.
  Progression is defined as:
  * ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement
  * Significant increase in T2 or fast fluid-attenuated inversion recovery (FLAIR) non-enhancing lesions on stable or increasing doses of corticosteroids
  * Any new lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor
  * Failure to return for evaluation as a result of death or deteriorating condition
  * Clear progression of non-measurable disease
Time Frame: From first dose to up to 6 months after first dose
Population: All treated participants in Cohorts 2-5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Percentage of participants | 9.4 [0.7 to 31.8] | 14.3 [2.3 to 36.6] | 0 [NA to NA] — Insufficient number of participants with events. | 20.0 [4.9 to 42.4] | 20.0 [3.1 to 47.5] | 11.4 [0.6 to 39.5] | 5.3 [0.4 to 21.4] | 14.0 [2.8 to 34.1]

10. Secondary Outcome: Overall Survival (OS), Cohorts 2-5
Description: Overall survival (OS) is defined as the time between date of first dose and the date of death for Cohorts 2-5.
Time Frame: From first dose to the date of death (up to approximately 55 months)
Population: All treated participants in Cohorts 2-5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Months | 6.67 [2.99 to 14.62] | 6.47 [2.14 to 13.17] | 7.36 [2.46 to 30.23] | 22.21 [13.77 to NA] — Insufficient number of participants with events. | 5.70 [1.81 to NA] — Insufficient number of participants with events. | 9.82 [2.50 to NA] — Insufficient number of participants with events.. | 5.91 [1.97 to 7.98] | 8.48 [3.45 to 17.28]

11. Secondary Outcome: Number of Treated Participants With Adverse Events (AEs)
Description: The number of treated participants who experienced an Adverse Event (AE) during the course of the study.
  An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Participants | 23 | 21 | 15 | 14 | 14 | 15 | 12 | 10 | 18 | 18

12. Secondary Outcome: Number of Treated Participants With Serious Adverse Events (SAEs)
Description: The number of treated participants who experienced a Serious Adverse Event (SAE) during the course of the study.
  SAE is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
  Note: The reporting timeframe of the SAEs for this Outcome Measure (first dose to 30 days post last dose) differs than that of the reporting timeframe of the SAEs reported under the AE section of the results form (first dose to 100 days post last dose) and thus, the data in each table of SAEs reflects the specific timeframe applied.
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Participants | 10 | 14 | 10 | 9 | 6 | 7 | 7 | 5 | 13 | 14

13. Secondary Outcome: Number of Treated Participants With Drug-Related Adverse Events
Description: The number of treated participants who experienced a Drug-Related Adverse Event during the course of the study.
  An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Participants | 14 | 16 | 12 | 8 | 6 | 11 | 6 | 6 | 11 | 10

14. Secondary Outcome: Number of Treated Participants With Adverse Events Leading to Discontinuation
Description: The number of treated participants who experienced an Adverse Event leading to discontinuation during the course of the study.
  An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Participants | 4 | 7 | 3 | 5 | 2 | 3 | 6 | 1 | 6 | 8

15. Secondary Outcome: Number of Treated Participant Deaths
Description: The number of treated participants who died during the course of the study.
Time Frame: From first dose to the date of death (up to approximately 55 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 22 | 16 | 15 | 15 | 15 | 12 | 10 | 19 | 19
Participants | 18 | 18 | 12 | 13 | 12 | 11 | 9 | 7 | 18 | 15

16. Secondary Outcome: Number of Treated Participant With Laboratory Abnormalities - Liver
Description: The number of treated participants who experienced a laboratory abnormality of the liver during the course of the study.
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN) Units per Liter (U/L) Results reported in International System of Units (SI)
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 23 | 21 | 16 | 12 | 13 | 14 | 11 | 10 | 19 | 18
Participants
  ALT OR AST > 3XULN | 3 | 7 | 2 | 0 | 0 | 3 | 1 | 1 | 3 | 2
  ALT OR AST > 5XULN | 2 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2
  ALT OR AST > 10XULN | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2
  ALT OR AST > 20XULN | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 23 | 21 | 15 | 12 | 13 | 14 | 11 | 10 | 19 | 18
  TOTAL BILIRUBIN > 2XULN | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ALP > 1.5XULN: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  ALP > 1.5XULN | 0 | 0 | 0 |  |  |  |  |  | 0 | 1
  ALT or AST > 3xULN w/ Tbili > 1.5*ULN within 1 day: number analyzed (Participants) | 23 | 21 | 15 | 12 | 13 | 14 | 11 | 10 | 19 | 18
  ALT or AST > 3xULN w/ Tbili > 1.5*ULN within 1 day | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT or AST > 3xULN w/ Tbili > 1.5*ULN within 30 days: number analyzed (Participants) | 23 | 21 | 15 | 12 | 13 | 14 | 11 | 10 | 19 | 18
  ALT or AST > 3xULN w/ Tbili > 1.5*ULN within 30 days | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT or AST > 3xULN w/ Tbili > 2*ULN within 1 day: number analyzed (Participants) | 23 | 21 | 15 | 12 | 13 | 14 | 11 | 10 | 19 | 18
  ALT or AST > 3xULN w/ Tbili > 2*ULN within 1 day | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT or AST > 3xULN w/ Tbili > 2*ULN within 30 days: number analyzed (Participants) | 23 | 21 | 15 | 12 | 13 | 14 | 11 | 10 | 19 | 18
  ALT or AST > 3xULN w/ Tbili > 2*ULN within 30 days | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

17. Secondary Outcome: Number of Treated Participant With Laboratory Abnormalities - Thyroid
Description: The number of treated participants who experienced a laboratory abnormality of the thyroid during the course of the study.
  Free T3 (FT3) Free T4 (FT4) Thyroid stimulating hormone (TSH) Lower Limit of Normal (LLN) Upper limit of normal (ULN) Milliunits per Liter (mlU/L) Results reported in International System of Units (SI)
Time Frame: From first dose to 30 days post-last dose (up to approximately an average of 3 months and a maximum of 51 months)
Population: All treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
Number analyzed (Participants) | 20 | 20 | 10 | 8 | 8 | 13 | 9 | 8 | 11 | 14
Participants
  TSH > ULN | 2 | 1 | 3 | 1 | 3 | 7 | 2 | 3 | 1 | 5
  TSH > ULN, WITH TSH <= ULN AT BASELINE | 2 | 1 | 2 | 1 | 0 | 7 | 1 | 3 | 1 | 2
  TSH > ULN, WITH AT LEAST ONE FT3/FT4 TEST < LLN | 1 | 1 | 1 | 1 | 1 | 6 | 2 | 2 | 0 | 2
  TSH > ULN, WITH ALL OTHER FT3/FT4 TEST >= LLN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  TSH > ULN, WITH FT3/FT4 TEST MISSING | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  TSH < LLN | 3 | 7 | 2 | 2 | 0 | 3 | 0 | 0 | 0 | 1
  TSH < LLN, WITH TSH >= LLN AT BASELINE | 3 | 6 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
  TSH<LLN, LLN WITH AT LEAST ONE FT3/FT4 TEST>ULN | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  TSH < LLN, WITH ALL OTHER FT3/FT4 TEST <= ULN | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
  TSH < LLN, WITH FT3/FT4 TEST MISSING | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Post Hoc Outcome: Overall Survival (OS), Cohort 1 Only - Extended Collection
Description: Overall survival (OS) is defined as the time between the date of diagnosis and the date of death in Cohort 1. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 17-Jan-2022).
Time Frame: From first dose to the date of death (up to approximately 55 months)
Population: All treated participants in Cohort 1
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Arm A1 | Arm B1
Number analyzed (Participants) | 23 | 22
Months | 11.66 [10.32 to 23.49] | 10.78 [9.13 to 15.77]

19. Post Hoc Outcome: Progression-Free Survival (PFS), Cohorts 2-4 - Extended Collection
Description: Progression-free survival (PFS) is defined as the time from first dose to the date of the first documented tumor progression or death due to any cause. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 17-Jan-2022).
  Progression is defined as:
  * ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement
  * Significant increase in T2 or fast fluid-attenuated inversion recovery (FLAIR) non-enhancing lesions on stable or increasing doses of corticosteroids
  * Any new lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor
  * Failure to return for evaluation as a result of death or deteriorating condition
  * Clear progression of non-measurable disease
Time Frame: as for outcome 7
Population: All treated participants in Cohorts 2-4
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 12 | 10
Months | 1.74 [1.35 to 2.73] | 1.38 [1.22 to 1.48] | 1.38 [1.22 to 1.38] | 2.69 [1.48 to 4.53] | 1.41 [1.38 to 2.60] | 4.60 [1.41 to 5.39]

20. Post Hoc Outcome: Progression-Free Survival (PFS), Cohort 5 Only - Extended Collection
Description: as for outcome 19
Time Frame: as for outcome 7
Population: All treated participants in Cohort 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A5 | Arm B5
Number analyzed (Participants) | 19 | 19
Months | 1.22 [1.08 to 1.31] | 1.61 [1.31 to 3.45]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to approximately 55 months). SAEs and Other AEs were monitored from first dose to 100 days after last dose (up to an average of 5 months and to a maximum of 53 months).
Description: Note: The reporting timeframe of the below SAEs (first dose to 100 days post last dose) differs than that of the reporting timeframe of the SAEs reported under the Outcome Measures section of the results form (first dose to 30 days post last dose) and thus, the data in each table of SAEs reflects the specific timeframe applied.
Arm/Group | Arm A1 | Arm B1 | Arm A2 | Arm B2 | Arm A3 | Arm B3 | Arm A4 | Arm B4 | Arm A5 | Arm B5
All-Cause Mortality (participants affected / at risk) | 18/23 | 18/22 | 12/16 | 13/15 | 12/15 | 11/15 | 9/12 | 7/10 | 18/19 | 15/19
Serious Adverse Events (participants affected / at risk) | 17/23 | 16/22 | 13/16 | 12/15 | 7/15 | 10/15 | 11/12 | 6/10 | 14/19 | 15/19
Other Adverse Events (participants affected / at risk) | 22/23 | 21/22 | 15/16 | 14/15 | 14/15 | 14/15 | 11/12 | 10/10 | 18/19 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1 (N=23) | Arm B1 (N=22) | Arm A2 (N=16) | Arm B2 (N=15) | Arm A3 (N=15) | Arm B3 (N=15) | Arm A4 (N=12) | Arm B4 (N=10) | Arm A5 (N=19) | Arm B5 (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated adverse reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multisystem inflammatory syndrome in children (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Measles (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7 | 6 | 5 | 6 | 2 | 7 | 5 | 7 | 7
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 4 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder dysfunction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1 (N=23) | Arm B1 (N=22) | Arm A2 (N=16) | Arm B2 (N=15) | Arm A3 (N=15) | Arm B3 (N=15) | Arm A4 (N=12) | Arm B4 (N=10) | Arm A5 (N=19) | Arm B5 (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 3 | 3 | 3 | 2 | 0 | 5 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Von Willebrand's disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 2 | 0 | 2 | 2 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal epithelium defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pupillary reflex impaired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 2 | 1 | 2 | 3 | 1 | 0 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 5 | 5 | 0 | 3 | 1 | 2 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 4 | 4 | 4 | 3 | 3 | 2 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 4 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 4 | 4 | 4 | 1 | 3 | 4 | 1 | 3 | 5
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 11 | 7 | 4 | 4 | 3 | 5 | 4 | 8 | 10
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 3 | 0 | 2 | 3 | 0 | 3 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 6 | 4 | 3 | 2 | 4 | 2 | 1 | 5 | 4
Gait disturbance (General disorders) | 4 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 2
Pyrexia (General disorders) | 5 | 6 | 2 | 4 | 1 | 2 | 3 | 2 | 2 | 5
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 2 | 1 | 0 | 1 | 2 | 3 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stoma site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access site rash (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 6 | 2 | 3 | 2 | 4 | 1 | 1 | 4 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anion gap increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 2 | 2 | 1 | 5 | 1 | 1 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Blood lactate dehydrogenase decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal transit time increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 3 | 0
Mean cell volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 3 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 0 | 2 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin turgor decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroxine free increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 7 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 2
Weight increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 3 | 2
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 3 | 2 | 3 | 3 | 2 | 0 | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 3 | 0 | 1 | 1 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 6 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 4
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 3 | 1 | 1 | 0 | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 6 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Consciousness fluctuating (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 10 | 7 | 2 | 7 | 6 | 5 | 2 | 13 | 5
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2
Meningism (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 2 | 3
Somnolence (Nervous system disorders) | 3 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VIth nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 1
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phonophobia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 3 | 2 | 3 | 3 | 1 | 4 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1 | 0 | 3 | 2 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0 | 3 | 1 | 1 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bloody discharge (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03130959/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03130959/SAP_002.pdf